CLINICAL TRIAL: NCT00462826
Title: A Phase II Evaluation of VEGF-Trap (AFLIBERCEPT, NSC #724770, NCI-Supplied Agent) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: VEGF Trap in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00597; NCI-2009-00597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000540237; GOG-0229F (Other: Gynecologic Oncology Group); GOG-0229F (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — aflibercept

ARMS (1):
- Treatment (aflibercept) (Experimental): Patients receive VEGF Trap IV over 1 hour on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap

SUMMARY:
This phase II trial is studying the side effects and how well VEGF Trap works in treating patients with recurrent or persistent endometrial cancer. VEGF Trap may stop the growth of endometrial cancer by blocking blood flow to the tumor and by carrying tumor-killing substances directly to endometrial cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the activity of VEGF Trap in patients with recurrent or persistent endometrial cancer, in terms of the frequency of patients who have progression-free survival for at least 6 months after initiating therapy or have objective tumor response.

II. Determine the toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the duration of progression-free survival and overall survival of patients treated with this drug.

OUTLINE:

Patients receive VEGF Trap IV over 1 hour on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma, meeting both of the following criteria:

  * Recurrent or persistent disease
  * Refractory to curative therapy or established treatments
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Tumors within a previously irradiated field are designated as nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days after completion of radiotherapy
* Must have received one prior chemotherapeutic regimen for management of endometrial carcinoma (initial treatment may include high-dose therapy, consolidation therapy, or extended therapy administered after surgical or non-surgical assessment)
* Not a candidate for a higher priority GOG protocol
* No history or evidence of primary brain tumor or brain metastases
* GOG performance status (PS) 0-2 (patients who received 1 prior regimen) OR GOG PS 0-1 (patients who received 2 prior regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Urine protein:creatinine ratio < 1.0 OR urine protein < 1.0 g by 24-hour urine collection
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* PT/PTT/INR ≤ 1.5 times ULN

  * In-range INR (between 2 and 3) allowed if patient is on a stable dose of therapeutic warfarin
* QTc < 500 msec
* No evidence of serious ventricular arrhythmia

  * Ventricular tachycardia or ventricular fibrillation must be < 3 beats in a row
* LVEF normal

  * Ejection fraction ≥ 50% (for patients who received prior anthracycline, including doxorubicin hydrochloride and/or doxorubicin hydrochloride liposome)
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension, defined as systolic blood pressure (BP) > 140 mm Hg or diastolic BP > 90 mm Hg
  * Myocardial infarction or unstable angina within the past 6 months
  * NYHA class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2
  * Cerebrovascular accident (i.e., CVA or stroke), transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* No HIV positivity
* No neuropathy (sensory and motor) > grade 1
* No active infection requiring antibiotics
* No other invasive malignancies or any evidence of other cancer within the past 5 years except for nonmelanoma skin cancer
* No serious nonhealing wound, ulcer, or bone fracture
* No history of abdominal fistula or gastrointestinal perforation
* No history or evidence of seizures not controlled with standard medical therapy
* No intra-abdominal abscess within the past 28 days
* No active bleeding or pathologic conditions that carry a high risk of bleeding (e.g., bleeding disorder, coagulopathy, or tumor involving major vessels)
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No significant traumatic injury within the past 28 days
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Recovered from prior surgery
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy and recovered
* At least 1 week since prior hormonal therapy

  * Concurrent hormone replacement therapy allowed
* At least 3 weeks since any other prior therapy, including immunologic agents
* One additional prior cytotoxic regimen for management of recurrent or persistent endometrial cancer allowed

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior minor surgery, fine needle aspirates, or core biopsies
* No prior cancer treatment that would preclude study compliance
* No prior noncytotoxic chemotherapy for management of recurrent or persistent endometrial disease
* No prior VEGF Trap or other VEGF pathway-targeted therapy
* More than 5 years since prior radiotherapy to any portion of the abdominal cavity or pelvis except for the treatment of endometrial cancer

  * More than 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin

    * Patient must remain free of recurrent or metastatic disease
* More than 5 years since prior chemotherapy for any abdominal or pelvic tumor except for the treatment of endometrial cancer

  * More than 3 years since prior adjuvant chemotherapy for localized breast cancer

    * Patient must remain free of recurrent or metastatic disease
* Concurrent low-molecular weight heparin allowed for the prevention or treatment of venous thromboembolic disease if condition is considered clinically stable with treatment
* No other concurrent investigational agents
* No concurrent major surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — Gynecologic Oncology Group
Locations (67):
- United States (67):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Jupiter Medical Center, Jupiter, Florida
  - Florida Hospital, Orlando, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Radiation Oncology Center of Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Stony Brook University Medical Center, Stony Brook, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - M D Anderson Cancer Center, Houston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Coleman RL, Sill MW, Lankes HA, Fader AN, Finkler NJ, Hoffman JS, Rose PG, Sutton GP, Drescher CW, McMeekin DS, Hu W, Deavers M, Godwin AK, Alpaugh RK, Sood AK. A phase II evaluation of aflibercept in the treatment of recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Dec;127(3):538-43. doi: 10.1016/j.ygyno.2012.08.020. Epub 2012 Aug 23. PMID 22922531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued to the first stage of accrual from 11/5/2007 to 6/2/2008. Patients were accrued to the second stage between 4/6/2009 and 7/13/2009. They received 4 mg/kg IV of VEGF-Trap every two weeks. One cycle was 28 days.
Pre-assignment Details: Patients were required to have had one prior chemotherapeutic regimen for the treatment of endometrial carcinoma. Patients entering the study therefore were required to have either persistent or recurrent cancer that was measurable by RECIST.
Period: Overall Study
Arm/Group | Treatment (Aflibercept)
Started | 49
Completed | 44
Not Completed | 5
Not completed — Ineligible - second primary | 1
Not completed — Ineligible - wrong cell type | 1
Not completed — Ineligible - wrong primary | 2
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Number of Eligible and Evaluable Participants
Arm/Group | Treatment (Aflibercept)
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.4)
Age, Customized [Number; unit: participants]
  40-49 years | 3
  50-59 years | 13
  60-69 years | 15
  70-79 years | 12
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44
International Federation of Gynecology and Obstetrics (FIGO) Recurrent/Persistent Disease [Number; unit: participants] | 44
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 1
  Endometrioid Adenocarcinoma | 23
  Mucinous Adenocarcinoma | 1
  Mixed Epithelial Carcinoma | 6
  Carcinsarcoma, MMT | 1
  Serous Adenocarcinoma | 11
Reason Off Study Therapy [Number; unit: participants]
  Disease Progression | 25
  Refused Further Treatment | 1
  Toxicity as permitted | 14
  Death | 3
  Other | 1
Tumor Response [Number; unit: participants]
  Partial Response | 3
  Stable Disease | 14
  Increase Disease | 16
  Indeterminate | 11

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival
Description: Number of participants who survived progression-free for more than 6 months.
Time Frame: At 6 monthsEvery other cycle during treatment for the first 6 months.
Measure: Number; unit: participants
Arm/Group | Treatment (Aflibercept)
Number analyzed (Participants) | 44
participants | 18

2. Primary Outcome: Objective Tumor Response (RECIST 1.0)
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle during treatment for the first 6 months, then every 3 months thereafter; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease; up to 5 years.
Population: Eligible and evaluable patients
Measure: Number; unit: participants
Arm/Group | Treatment (Aflibercept)
Number analyzed (Participants) | 44
participants
  Complete Response | 0
  Partial Response | 3

3. Primary Outcome: Number of Participants With Incidence of Adverse Events at Least Possibly Related to Study Agent as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Adverse events at least possibly related to the study agent.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and evaluable patients.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 44 | 44 | 44 | 44 | 44 | 44
Participants
  Leukopenia | 37 | 7 | 0 | 0 | 0 | 0
  Thrombocytopenia | 36 | 5 | 2 | 1 | 0 | 0
  Neutropenia | 41 | 0 | 1 | 1 | 1 | 0
  Anemia | 25 | 9 | 9 | 1 | 0 | 0
  Other hematologic | 40 | 3 | 1 | 0 | 0 | 0
  Allergy/Immunology | 40 | 3 | 1 | 0 | 0 | 0
  Cardiac | 23 | 1 | 8 | 10 | 2 | 0
  Coagulation | 39 | 3 | 1 | 1 | 0 | 0
  Constitutional | 16 | 13 | 12 | 3 | 0 | 0
  Dermatologic | 36 | 6 | 2 | 0 | 0 | 0
  Endocrine | 42 | 2 | 0 | 0 | 0 | 0
  Nausea | 25 | 12 | 4 | 3 | 0 | 0
  Vomiting | 32 | 6 | 4 | 2 | 0 | 0
  Gastrointestinal | 14 | 15 | 10 | 3 | 1 | 1
  Genitourinary/renal | 41 | 2 | 0 | 1 | 0 | 0
  Hemorrhage | 36 | 5 | 0 | 1 | 2 | 0
  Infection | 39 | 0 | 3 | 2 | 0 | 0
  Lymphatics | 40 | 3 | 1 | 0 | 0 | 0
  Metabolic | 27 | 10 | 3 | 3 | 1 | 0
  Musculoskeletal | 41 | 2 | 0 | 1 | 0 | 0
  Neurosensory | 38 | 4 | 2 | 0 | 0 | 0
  Other neurological | 31 | 7 | 1 | 2 | 3 | 0
  Ocular/visual | 42 | 1 | 1 | 0 | 0 | 0
  Pain | 13 | 15 | 8 | 8 | 0 | 0
  Pulmonary | 23 | 13 | 4 | 3 | 1 | 0
  Vascular | 43 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Duration of Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Eligible and evaluable patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Aflibercept)
Number analyzed (Participants) | 44
months | 2.9 [2.1 to 6.21]

5. Secondary Outcome: Duration of Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and evaluable patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Aflibercept)
Number analyzed (Participants) | 44
months | 14.5 [9.86 to 20.44]

ADVERSE EVENTS:
Time Frame: From the time of study activation until 7-8-2011 when the last form was submitted.
Arm/Group | Treatment (Aflibercept)
Serious Adverse Events (participants affected / at risk) | 24/44
Other Adverse Events (participants affected / at risk) | 28/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Aflibercept) (N=44)
Neutrophils (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 2
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Fever (General disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 3
Perforation, Gi - Colon (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Hemorrhage, Cns (Vascular disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Cns Ischemia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Chest Wall (General disorders) | 1
Vascular - Other (Vascular disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Aflibercept) (N=44)
Rhinitis (Immune system disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 5
Platelets (Blood and lymphatic system disorders) | 9
Leukocytes (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 22
Hypertension (Cardiac disorders) | 19
Inr (Vascular disorders) | 3
Ptt (Vascular disorders) | 3
Weight Loss (General disorders) | 3
Fatigue (General disorders) | 28
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 6
Hot Flashes (Endocrine disorders) | 3
Dysphagia (Gastrointestinal disorders) | 5
Taste Alteration (Gastrointestinal disorders) | 3
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 3
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 12
Anorexia (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 19
Diarrhea (Gastrointestinal disorders) | 10
Hemorrhage, Gu - Vagina (Vascular disorders) | 3
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 5
Edema: Limb (Blood and lymphatic system disorders) | 5
Ast (Metabolism and nutrition disorders) | 9
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 3
Proteinuria (Metabolism and nutrition disorders) | 4
Creatinine (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Alt (Metabolism and nutrition disorders) | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 3
Mood Alteration - Depression (Nervous system disorders) | 9
Neuropathy-Sensory (Nervous system disorders) | 18
Blurred Vision (Eye disorders) | 3
Pain: Head/Headache (General disorders) | 17
Pain: Extremity-Limb (General disorders) | 5
Pain: Joint (General disorders) | 10
Pain: Abdominal Pain Nos (General disorders) | 9
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Urinary Frequency (Renal and urinary disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less